CLINICAL TRIAL: NCT01238822
Title: Response Variability in Children With ADHD
Brief Title: Response Variability in Children With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: R01MH074770 (NIH)
Record Dates: First submitted 2010-11-09; First posted 2010-11-11 (Estimated); Results first posted 2012-04-04 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo
- Low Dose Methylphenidate (Active Comparator): Low dose: 18 mg methylphenidate
  Interventions: Drug: Methylphenidate
- Medium Dose Methylphenidate (Active Comparator): Medium Dosage: 36 mg if more than 50 kg and 27 mg if less than 50 kg
  Interventions: Drug: Methylphenidate
- High Dose Methylphenidate (Active Comparator): 54 mg if more than 50 kg and 36 mg if less than 50 kg
  Interventions: Drug: Methylphenidate

INTERVENTIONS:
Drug: Methylphenidate — 18 mg methylphenidate
  Other Names: Concerta
  Arms: Low Dose Methylphenidate
Drug: placebo — Placebo
  Arms: Placebo
Drug: Methylphenidate — 36 mg methylphenidate
  Other Names: Concerta
  Arms: Medium Dose Methylphenidate
Drug: Methylphenidate — 54 mg methylphenidate
  Other Names: Concerta
  Arms: High Dose Methylphenidate

SUMMARY:
Children with Attention Deficit Hyperactivity Disorder (ADHD) have numerous areas of neuropsychological dysfunction including response inhibition, working memory, and attention. One neuropsychological outcome measure that consistently reveals between-group differences is response variability. However, until recently, differences in response variability have been reported as an ancillary finding or viewed as a nuisance in the analyses. The specific aims of the present study are to 1) Examine response variability in ADHD patients across neuropsychological tasks to understand the breadth of this specific deficit and to understand the relation between response variability and other neuropsychological outcome measures; 2) Assess whether response variability deficits are specific to either or both of the two most prevalent ADHD subtypes (i.e., Combined Type [CT] and Predominantly Inattentive Type [PIT]); 3) Determine whether response variability in ADHD patients is affected by either medication or a variety of environmental manipulations (e.g., reward); and 4) Understand the relationship between neuropsychological measures of response variability and naturalistic instances of variable performance. Forty-five children (aged 7-11) with ADHD-CT, 45 children with ADHD-PIT, and 45 normal controls will be recruited to examine response variability across a wide range of neuropsychological tests. Task parameters such as event rate, stimulus saliency, and the presence of operant reward will be modified on each test to determine the conditions under which response variability is manifested in children with ADHD. In addition, all children with ADHD will participate in a placebo-controlled, randomized medication trial with a psychostimulant medication to assess the effects of medication on response variability. Advanced analytic methods utilizing non-Gaussian distributions and fast Fourier Transforms of the reaction time data will be used to conduct detailed analyses of RT patterns across the ADHD and normal control groups. Further, the effects of task parametric manipulations and medication on response variability will be examined. Finally, relations between response variability on neuropsychological tests and response variability in a variety of real-world analog situations will be examined to evaluate the ecological validity of these deficits.

ELIGIBILITY:
Inclusion Criteria. Participants for the study must meet all of the following criteria:

1. Consent: The family must provide signature of informed consent by parents or legal guardians.
2. Age at time of Screening: 7 years to 11 years, inclusive
3. Gender: includes male and female children.
4. ADHD Diagnostic Status: ADHD patients must meet DSM-IV criteria for ADHD, Inattentive or Combined subtype. Normal controls must not meet DSM-IV criteria for ADHD, any subtype. Section D.4 below describes in detail the diagnostic process for arriving at diagnosis.
5. Cognitive Functioning: IQ of greater than 80 as estimated by Vocabulary and Block Design subtests of the Wechsler Intelligence Scale for Children, Fourth Edition (WISC-IV).
6. Learning Disability: All children will be administered the abbreviated WIAT including the Spelling, Reading, and Math subtests. Children must score above 80 on all three WIAT subtests.
7. School: Children must be enrolled in a school setting from which teacher ratings can be obtained.

Exclusion Criteria. Potential participants will be excluded if they meet any of the following criteria:

1. Understanding Level. The patient and parent cannot understand or follow instructions given in the study.
2. History of Psychiatric Medications: Children who have a history of taking any medication for psychological or psychiatric problems will be excluded from participation.
3. Exclusionary Psychiatric Conditions: Children whose primary diagnosis is something other than ADHD will be excluded from participation.
4. Developmental Disabilities. As a result of scores on the IQ screening, additional assessments, or the judgment of the study clinicians, patients will be excluded if they are deemed to be significantly developmentally delayed. This includes clinically significant delays in cognitive function or the presence of other Pervasive Developmental Disorders (PDD).
5. Organic Brain Injury: Children must not have a history of head trauma, neurological disorder, or any other organic disorder that could possibly affect brain function.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2006-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Childrens Hospital, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Froehlich TE, Epstein JN, Nick TG, Melguizo Castro MS, Stein MA, Brinkman WB, Graham AJ, Langberg JM, Kahn RS. Pharmacogenetic predictors of methylphenidate dose-response in attention-deficit/hyperactivity disorder. J Am Acad Child Adolesc Psychiatry. 2011 Nov;50(11):1129-1139.e2. doi: 10.1016/j.jaac.2011.08.002. Epub 2011 Sep 15. PMID 22024001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children were recruited through multiple community and clinical sources including schools and local practitioners to participate in a study of the effects of medication on cognitive functioning. Diagnostic status was determined using methodology similar to that employed by the Multimodal Treatment Study of ADHD (MTA Cooperative Group, 1999).
Groups:
- All Participants: All participants received 3 weekly doses of methylphenidate at a low dose (18 mg), medium dosage (27 mg or 36 mg depending on weight) and a high dosage (52 mg or 36 mg depending on weight) and another week of placebo. Patients took each dosage for 1 week and parents and teachers rated their behavior at the end of each week.
Period: Overall Study
Arm/Group | All Participants
Started | 96
Received Placebo | 93
Received Low Dosage | 93
Received Medium Dosage | 93
Received High Dosage | 93
Completed | 93
Not Completed | 3
Not completed — COULD NOT SWALLOW PILLS | 3

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 96
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 8.11 (1.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 70
Region of Enrollment [Number; unit: participants]
  United States | 96

OUTCOME MEASURES:

1. Primary Outcome: Attention Deficit / Hyperactivity Disorder Total Sum Score of All 18 ADHD Symptom Items
Description: Parent and teacher Vanderbilt ADHD Rating Scales - Attention Deficit / Hyperactivity Disorder Total sum score of all 18 ADHD symptom items - range equals 0-54
  O - No ADHD symptoms 54 - Highest ADHD symptoms
Time Frame: end of first week, end of second week, end of third week, end of fourth week. Total of 4 weeks.
Population: Intent to treat with imputation for missing data.
Measure: Mean (Standard Deviation); unit: Score
Groups:
- Low Dosage: 18 mg methylphenidate
- Medium Dosage: 36 mg methylphenidate if >25 kg; 27 mg methylphenidate if < 25 kg.
- High Dosage: 54 mg methylphenidate if >25 kg; 36 mg methylphenidate if < 25 kg.
Arm/Group | Placebo | Low Dosage | Medium Dosage | High Dosage
Number analyzed (Participants) | 96 | 96 | 96 | 96
Score | 26.54 (12.03) | 25 (12.73) | 18.94 (11.18) | 18.46 (11.68)

ADVERSE EVENTS:
Groups:
- Low Dosage: Low dose: 18 mg methylphenidate
- Medium Dosage: Medium Dosage: 36 mg methylphenidate
- High Dosage: 54 mg methylphenidate
Arm/Group | Placebo | Low Dosage | Medium Dosage | High Dosage
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/96 | 1/96 | 0/96
Other Adverse Events (participants affected / at risk) | 13/96 | 12/96 | 16/96 | 37/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=96) | Low Dosage (N=96) | Medium Dosage (N=96) | High Dosage (N=96)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=96) | Low Dosage (N=96) | Medium Dosage (N=96) | High Dosage (N=96)
Parent reported tics (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) — Number rated 4 (severe)
Parent-reported buccal-lingual movements (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) — Number rated 4 (severe)
Parent-reported picking at skin or fingers, nail-biting, or cheek chewing (Nervous system disorders) | 3 (3) | 1 (1) | 3 (3) | 7 (7) — Number rated 4 (severe)
Parent-reported worried/anxious (Psychiatric disorders) | 2 (2) | 3 (3) | 5 (5) | 9 (9) — Number rated 4 (severe)
Parent-reported dull, tired, listless (Nervous system disorders) | 4 (4) | 3 (3) | 2 (2) | 7 (7) — Number rated 4 (severe)
Parent-reported headaches (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Number rated 4 (severe)
Parent-reported stomachache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Number rated 4 (severe)
Parent-reported crabby, irritable (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Number rated 4 (severe)
Parent-reported tearful, sad, depressed (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Number rated 4 (severe)
Parent-reported socially withdrawn (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) — Number rated 4 (severe)
Parent-reported hallucinations (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) — Number rated 4 (severe)
Parent-reported loss of appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) — Number rated 4 (severe)
Parent-reported trouble sleeping (Psychiatric disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) — Number rated 4 (severe)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No